CLINICAL TRIAL: NCT03817476
Title: Relative Bioavailability of Batch 1 and Batch 2 of the Intended Commercial Formulation of BI 425809 Compared to Each Other and to TF 2 Formulation of BI 425809 Following Oral Administration in Healthy Male and Female Subjects (Randomized, Open-label, Single-dose, Three-treatment, Three-period, Six-sequence Crossover Study)
Brief Title: A Study in Healthy People to Test if Taking Different Formulations of BI 425809 Tablets Influences the Amount of BI 425809 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0019; 2018-003625-29 (EudraCT Number)
Record Dates: First submitted 2019-01-24; First posted 2019-01-25 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Healthy
MeSH Terms: interventions — BI 425809

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- T1-T2-R (Experimental)
  Interventions: Drug: BI 425809 (Treatment T1); Drug: BI 425809 (Treatment T2); Drug: BI 425809 (Treatment R)
- T1-R-T2 (Experimental)
  Interventions: Drug: BI 425809 (Treatment T1); Drug: BI 425809 (Treatment T2); Drug: BI 425809 (Treatment R)
- T2-T1-R (Experimental)
  Interventions: Drug: BI 425809 (Treatment T1); Drug: BI 425809 (Treatment T2); Drug: BI 425809 (Treatment R)
- T2-R-T1 (Experimental)
  Interventions: Drug: BI 425809 (Treatment T1); Drug: BI 425809 (Treatment T2); Drug: BI 425809 (Treatment R)
- R-T1-T2 (Experimental)
  Interventions: Drug: BI 425809 (Treatment T1); Drug: BI 425809 (Treatment T2); Drug: BI 425809 (Treatment R)
- R-T2-T1 (Experimental)
  Interventions: Drug: BI 425809 (Treatment T1); Drug: BI 425809 (Treatment T2); Drug: BI 425809 (Treatment R)

INTERVENTIONS:
Drug: BI 425809 (Treatment T1) — Intended commercial formulation tablet from batch 1 (iCF1)
Drug: BI 425809 (Treatment T2) — Intended commercial formulation tablet from batch 2 (iCF2)
Drug: BI 425809 (Treatment R) — Trial formulation 2 tablet (TF2)

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of batch 1 of the intended commercial tablet formulation (iCF1) of BI 425809 vs batch 2 of the intended commercial tablet formulation (iCF2) of BI 425809 vs BI 425809 (TF2) formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation
* Male subjects, or female subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods plus condom:

    --- implants, injectables, combined oral or vaginal contraceptives, intrauterine device
  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant Electrocardiogram (ECG) finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Female subjects, only: Positive pregnancy test, pregnancy, or plans to become pregnant within 30 days after study completion
* Female subjects, only: Lactation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
AUC0-72 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 72 h) | Up to 72 hours
Cmax (maximum measured concentration of the analyte in plasma) | Up to 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/